CLINICAL TRIAL: NCT05939063
Title: Laparoscopic Radical Antegrade Modular Pancreatosplenectomy Versus Laparoscopic Distal Pancreatosplecnectomy in Selected Left-sided Pancreatic Cancer: a Multicenter Randomized Controlled Clinical Trial
Brief Title: LRAMPS Versus LDP in Selected Early-stage Left-sided Pancreatic Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: The Third Affiliated Hospital of Soochow University (Other); Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, President of Fudan University Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPAC-6
Record Dates: First submitted 2023-07-02; First posted 2023-07-11 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Left-sided Pancreatic Cancer
Keywords: Left-sided pancreatic cancer; Early-stage tumor; Laparoscopic radical antegrade modular pancreatosplenectomy; Laparoscopic distal pancreatosplecnectomy; Surgical complication; Oncologic prognosis
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LRAMPS group (Active Comparator): Patients who meet the inclusion and exclusion criteria will undergo laparoscopic radical antegrade modular pancreatosplenectomy (LRAMPS) surgery.
  Interventions: Procedure: LRAMPS
- LDP group (Experimental): Patients who meet the inclusion and exclusion criteria will undergo laparoscopic distal pancreatosplecnectomy (LDP) surgery.
  Interventions: Procedure: LDP

INTERVENTIONS:
Procedure: LRAMPS — For LRAMPS procedure, Gerota's fascia and perirenal fat capsule are removed, and the procedure is divided into anterior LRAMPS and posterior LRAMPS depending on whether the left adrenal gland is resected. The N1 station lymph nodes (i.e., groups 10, 11, and 18) in the body and tail of the pancreas are removed. If the tumor is located near the pancreatic body, the No. 9 lymph node group is additionally removed.
  Arms: LRAMPS group
Procedure: LDP — For LDP procedure, the dissection plane is located behind the fusion fascia. The N1 station lymph nodes (i.e., groups 10, 11, and 18) in the body and tail of the pancreas are removed. If the tumor is located near the pancreatic body, the No. 9 lymph node group is additionally removed.
  Arms: LDP group

SUMMARY:
This multicenter randomized controlled clinical trial proposed the criteria for selecting patients with early-stage left-sided pancreatic cancer and aimed to compare the perioperative and oncological outcomes of patients within the criteria who underwent laparoscopic radical antegrade modular pancreatosplenectomy versus laparoscopic distal pancreatosplenectomy.

DETAILED DESCRIPTION:
Although prospective comparative studies are lacking, laparoscopic distal pancreatosplenectomy (LDP) was considered to be feasible, safe, and oncologically equivalent for treating pancreatic ductal adenocarcinoma (PDAC). However, the extent of posterior resection and the oncological safety of achieving complete N1 lymph node resection in LDP remain uncertain. Strasberg proposed radical antegrade modular pancreatosplenectomy (RAMPS) for the treatment of resectable left-sided PDAC and confirmed that this technique can achieve negative margins and satisfactory survival. Given the oncological equivalence of laparoscopic radical antegrade modular pancreatosplenectomy (LRAMPS) and its advantages in short-term outcomes, several studies have assessed the feasibility of LRAMPS as the standard treatment for resectable left-sided PDAC. However, previous studies on LRAMPS have mostly included tumors staged T2 and above, and there is currently no research on the routine use of LRAMPS for early-stage tumors. We proposed the criteria for selecting patients with early-stage left-sided PDAC: (1) diameter ≤ 4 cm; (2) located ≥ 1 cm from the celiac trunk; (3) didn't invade the fascial layer behind the pancreas. This multicenter open-label randomized controlled clinical trial aims to compare the perioperative and oncological outcomes of patients within the criteria who underwent LRAMPS versus LDP.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed as resectable left-sided pancreatic cancer before surgery.
* Imaging tumor diameter ≤ 4 cm.
* Located ≥ 1cm from the celiac trunk.
* Tumor didn't invade the fascial layer behind the pancreas.
* Be able to comply with research protocol.
* Voluntary participation and signed informed consent.

Exclusion Criteria:

* Received neoadjuvant therapy.
* Presence of liver or other distant metastasis.
* Multifocal or recurrent disease.
* History of other malignancies.
* Simultaneously participating in other clinical trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
R0 retroperitoneal margin rate | From the date of surgery to 1 month after surgery.
  R0 retroperitoneal margin rate diagnosed by postoperative pathological examination.
R0 transection margin rate | From the date of surgery to 1 month after surgery.
  R0 transection margin rate diagnosed by postoperative pathological examination.
Lymph node positive rate | From the date of surgery to 1 month after surgery.
  Lymph node positive rate diagnosed by postoperative pathological examination.

SECONDARY OUTCOMES:
Perioperative complication rate | Within 90 days after surgery.
  Adverse events that occur during or after the surgery, including the incidence of postoperative complications reported according to the Clavien-Dindo classification, clinical relevant postoperative pancreatic fistula (POPF), postoperative pancreatic hemorrhage (PPH), delayed gastric emptying (DGE), reoperation rate and mortality rate within 90 days after surgery.
Life quality satisfaction evaluated according to EORTC C30 scale | Through study completion, an average of 3 year.
  The patient's health-related quality of life after surgical intervention. It includes physical, emotional, and social aspects of a patient's well-being. This study evaluated quality of life using a telephone survey and the EORTC C30 scales.
Recurrence-free survival (RFS) | Through study completion, an average of 3 year.
  The time of surgery to the time of tumor recurrence or death.
Overall survival (OS) | Through study completion, an average of 3 year.
  The time from the surgery to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Xianjun Yu, MD, PhD, Principal Investigator — Fudan University; Xiaowu Xu, MD, Study Director — Fudan University
Locations (1):
- Department of Pancreatic Surgery, Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Rooij T, van Hilst J, van Santvoort H, Boerma D, van den Boezem P, Daams F, van Dam R, Dejong C, van Duyn E, Dijkgraaf M, van Eijck C, Festen S, Gerhards M, Groot Koerkamp B, de Hingh I, Kazemier G, Klaase J, de Kleine R, van Laarhoven C, Luyer M, Patijn G, Steenvoorde P, Suker M, Abu Hilal M, Busch O, Besselink M; Dutch Pancreatic Cancer Group. Minimally Invasive Versus Open Distal Pancreatectomy (LEOPARD): A Multicenter Patient-blinded Randomized Controlled Trial. Ann Surg. 2019 Jan;269(1):2-9. doi: 10.1097/SLA.0000000000002979. PMID 30080726
- [Background] Asbun HJ, Moekotte AL, Vissers FL, Kunzler F, Cipriani F, Alseidi A, D'Angelica MI, Balduzzi A, Bassi C, Bjornsson B, Boggi U, Callery MP, Del Chiaro M, Coimbra FJ, Conrad C, Cook A, Coppola A, Dervenis C, Dokmak S, Edil BH, Edwin B, Giulianotti PC, Han HS, Hansen PD, van der Heijde N, van Hilst J, Hester CA, Hogg ME, Jarufe N, Jeyarajah DR, Keck T, Kim SC, Khatkov IE, Kokudo N, Kooby DA, Korrel M, de Leon FJ, Lluis N, Lof S, Machado MA, Demartines N, Martinie JB, Merchant NB, Molenaar IQ, Moravek C, Mou YP, Nakamura M, Nealon WH, Palanivelu C, Pessaux P, Pitt HA, Polanco PM, Primrose JN, Rawashdeh A, Sanford DE, Senthilnathan P, Shrikhande SV, Stauffer JA, Takaori K, Talamonti MS, Tang CN, Vollmer CM, Wakabayashi G, Walsh RM, Wang SE, Zinner MJ, Wolfgang CL, Zureikat AH, Zwart MJ, Conlon KC, Kendrick ML, Zeh HJ, Hilal MA, Besselink MG; International Study Group on Minimally Invasive Pancreas Surgery (I-MIPS). The Miami International Evidence-based Guidelines on Minimally Invasive Pancreas Resection. Ann Surg. 2020 Jan;271(1):1-14. doi: 10.1097/SLA.0000000000003590. PMID 31567509
- [Background] van Hilst J, de Rooij T, Klompmaker S, Rawashdeh M, Aleotti F, Al-Sarireh B, Alseidi A, Ateeb Z, Balzano G, Berrevoet F, Bjornsson B, Boggi U, Busch OR, Butturini G, Casadei R, Del Chiaro M, Chikhladze S, Cipriani F, van Dam R, Damoli I, van Dieren S, Dokmak S, Edwin B, van Eijck C, Fabre JM, Falconi M, Farges O, Fernandez-Cruz L, Forgione A, Frigerio I, Fuks D, Gavazzi F, Gayet B, Giardino A, Groot Koerkamp B, Hackert T, Hassenpflug M, Kabir I, Keck T, Khatkov I, Kusar M, Lombardo C, Marchegiani G, Marshall R, Menon KV, Montorsi M, Orville M, de Pastena M, Pietrabissa A, Poves I, Primrose J, Pugliese R, Ricci C, Roberts K, Rosok B, Sahakyan MA, Sanchez-Cabus S, Sandstrom P, Scovel L, Solaini L, Soonawalla Z, Souche FR, Sutcliffe RP, Tiberio GA, Tomazic A, Troisi R, Wellner U, White S, Wittel UA, Zerbi A, Bassi C, Besselink MG, Abu Hilal M; European Consortium on Minimally Invasive Pancreatic Surgery (E-MIPS). Minimally Invasive versus Open Distal Pancreatectomy for Ductal Adenocarcinoma (DIPLOMA): A Pan-European Propensity Score Matched Study. Ann Surg. 2019 Jan;269(1):10-17. doi: 10.1097/SLA.0000000000002561. PMID 29099399
- [Background] Strasberg SM, Drebin JA, Linehan D. Radical antegrade modular pancreatosplenectomy. Surgery. 2003 May;133(5):521-7. doi: 10.1067/msy.2003.146. PMID 12773980
- [Background] Strasberg SM, Linehan DC, Hawkins WG. Radical antegrade modular pancreatosplenectomy procedure for adenocarcinoma of the body and tail of the pancreas: ability to obtain negative tangential margins. J Am Coll Surg. 2007 Feb;204(2):244-9. doi: 10.1016/j.jamcollsurg.2006.11.002. Epub 2007 Jan 4. PMID 17254928
- [Background] Mitchem JB, Hamilton N, Gao F, Hawkins WG, Linehan DC, Strasberg SM. Long-term results of resection of adenocarcinoma of the body and tail of the pancreas using radical antegrade modular pancreatosplenectomy procedure. J Am Coll Surg. 2012 Jan;214(1):46-52. doi: 10.1016/j.jamcollsurg.2011.10.008. PMID 22192922
- [Background] Takahashi A, Mise Y, Watanabe G, Yoshioka R, Ono Y, Inoue Y, Ito H, Takahashi Y, Kawasaki S, Saiura A. Radical antegrade modular pancreatosplenectomy enhances local control of the disease in patients with left-sided pancreatic cancer. HPB (Oxford). 2023 Jan;25(1):37-44. doi: 10.1016/j.hpb.2022.08.004. Epub 2022 Aug 20. PMID 36088222
- [Background] Tang W, Zhang YF, Zhao YF, Wei XF, Xiao H, Wu Q, Du CY, Qiu JG. Comparison of laparoscopic versus open radical antegrade modular pancreatosplenectomy for pancreatic cancer: A systematic review and meta-analysis. Int J Surg. 2022 Jul;103:106676. doi: 10.1016/j.ijsu.2022.106676. Epub 2022 May 13. PMID 35577311
- [Background] Zhang H, Li Y, Liao Q, Xing C, Ding C, Zhang T, Guo J, Han X, Xu Q, Wu W, Zhao Y, Dai M. Comparison of minimal invasive versus open radical antegrade modular pancreatosplenectomy (RAMPS) for pancreatic ductal adenocarcinoma: a single center retrospective study. Surg Endosc. 2021 Jul;35(7):3763-3773. doi: 10.1007/s00464-020-07938-1. Epub 2020 Oct 8. PMID 33033915
- [Background] Wu EJ, Kabir T, Zhao JJ, Goh BKP. Minimally Invasive Versus Open Radical Antegrade Modular Pancreatosplenectomy: A Meta-Analysis. World J Surg. 2022 Jan;46(1):235-245. doi: 10.1007/s00268-021-06328-5. Epub 2021 Oct 5. PMID 34609574
- [Background] Lee SH, Kang CM, Hwang HK, Choi SH, Lee WJ, Chi HS. Minimally invasive RAMPS in well-selected left-sided pancreatic cancer within Yonsei criteria: long-term (>median 3 years) oncologic outcomes. Surg Endosc. 2014 Oct;28(10):2848-55. doi: 10.1007/s00464-014-3537-3. Epub 2014 May 23. PMID 24853839
- [Background] Sato S, Oba A, Kato T, Kobayashi K, Wu YHA, Ono Y, Sato T, Ito H, Inoue Y, Takahashi Y. Feasibility of laparoscopic radical antegrade modular pancreatosplenectomy (RAMPS) as a standard treatment for distal resectable pancreatic cancer. Langenbecks Arch Surg. 2023 May 30;408(1):217. doi: 10.1007/s00423-023-02942-0. PMID 37249638
- [Background] Sutton TL, Potter KC, Mayo SC, Pommier R, Gilbert EW, Sheppard BC. Complications in Distal Pancreatectomy versus Radical Antegrade Modular Pancreatosplenectomy: A Disease Risk Score Analysis Utilizing National Surgical Quality Improvement Project Data. World J Surg. 2022 Jul;46(7):1768-1775. doi: 10.1007/s00268-022-06545-6. Epub 2022 Apr 11. PMID 35403874
- [Background] Sivasanker M, Desouza A, Bhandare M, Chaudhari V, Goel M, Shrikhande SV. Radical antegrade modular pancreatosplenectomy for all pancreatic body and tail tumors: rationale and results. Langenbecks Arch Surg. 2019 Mar;404(2):183-190. doi: 10.1007/s00423-019-01763-4. Epub 2019 Feb 21. PMID 30790046